CLINICAL TRIAL: NCT06665555
Title: A Phase 1, Open-label Study to Evaluate the Safety and Plasma and Intrapulmonary Pharmacokinetics of Ceftibuten and Ledaborbactam in Healthy Adult Participants
Brief Title: Plasma and Intrapulmonary Pharmacokinetics of Ceftibuten and Ledaborbactam in Healthy Male and Female Participants 18 to ≤55 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VNRX-7145-105
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetics; Healthy Volunteers
MeSH Terms: interventions — Ceftibuten

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants in Group 1 will undergo one standardized bronchoscopy with bronchoalveolar lavage after the fifth dose of ceftibuten-ledaborbactam etzadroxil.
  Interventions: Drug: ledaborbactam etzadroxil; Drug: ceftibuten
- Group 2 (Experimental): Participants in Group 2 will undergo one standardized bronchoscopy with bronchoalveolar lavage after the fifth of dose of ceftibuten alone.
  Interventions: Drug: ceftibuten

INTERVENTIONS:
Drug: ledaborbactam etzadroxil — Five doses of ledaborbactam etzadroxil will be administered orally every 12 hours
  Arms: Group 1
Drug: ceftibuten — Five doses of ceftibuten will be administered orally every 12 hours

SUMMARY:
This is a Phase 1, open-label, single-center PK study in healthy adult male and female participants between 18 and 55 years of age (both inclusive). Thirty-one participants will each undergo one standard bronchoscopy with bronchoalveolar lavage (BAL) following the fifth dose of ceftibuten-ledaborbactam etzadroxil or ceftibuten alone. BAL fluid samples and plasma samples will be collected at designated timepoints to determine the concentrations of ceftibuten, ledaborbactam, and urea.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-55 years
* Males or non-pregnant, non-lactating females
* Body Mass Index: ≥18 and ≤32 kg/m2
* Forced expiratory volume in 1 second of at least 80% of predicted value
* Laboratory values meeting defined entry criteria

Exclusion Criteria:

* History of drug allergy or hypersensitivity to penicillin, cephalosporin, or β-lactam antibacterial drug or to medications used during a bronchoscopy
* Conditions that potentially alter absorption and/or excretion of orally administered drugs
* History or presence of significant diseases, including any clinically relevant acute illness or surgery within the past 3 months
* Positive alcohol, drug, or tobacco use/test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Intrapulmonary PK - AUC0-12 (ceftibuten) | 0-12 hours after 5th dose
  Area under the curve from time zero to 12 hours
Intrapulmonary PK - AUC0-12 (ledaborbactam) | 0-12 hours after 5th dose
  Area under the curve from time zero to 12 hours
Plasma PK - Cmax (ceftibuten) | 0-12 hours after 5th dose
  Maximum concentration
Plasma PK - Cmax (ledaborbactam) | 0-12 hours after 5th dose
  Maximum concentration
Plasma PK - AUC0-12 (ceftibuten) | Time Frame: 0-12 hours after 5th dose
  Area under the curve from time zero to 12 hours
Plasma PK - AUC0-12 (ledaborbactam) | 0-12 hours after 5th dose
  Area under the curve from time zero to 12 hours
Ratios of drug exposure in ELF to plasma using the AUC values for each matrix | 0-12 hours after 5th dose

SECONDARY OUTCOMES:
Proportion of participants experiencing treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Day 1 - Day 8
Proportion of participants discontinuing study drug due to TEAEs and SAEs | Day 1 - Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hamed, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- Pulmonary Associates, Phoenix, Arizona, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-12-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT06665555/ICF_000.pdf